CLINICAL TRIAL: NCT05079321
Title: Ocular Effects of Scleral Lens Wear on Dry Eye Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 40887
Record Dates: First submitted 2021-10-01; First posted 2021-10-15 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2023-11

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Coated Scleral Lens (Experimental): Participants wear a lens coated with Hydra-PEG.
  Interventions: Device: Hydra-PEG
- Uncoated Scleral Lens (Placebo Comparator): Participants wear an uncoated (control) lens.
  Interventions: Device: Uncoated

INTERVENTIONS:
Device: Hydra-PEG — Zen™ RC scleral lenses (Hydra-PEG coated)
  Arms: Coated Scleral Lens
Device: Uncoated — Zen™ RC scleral lenses (non-coated)
  Arms: Uncoated Scleral Lens

SUMMARY:
The purpose of this study is to investigate the effects of scleral contact lens wear on a DE population using coated (Hydra-PEG) and uncoated (control) lenses. Symptoms of DE, quality of the tear film, quality of life, epithelial and overall corneal thickness, vision and comfort will be assessed before and after dispensing and wearing the lenses for four weeks.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

* Is at least 18 years of age and has full legal capacity to volunteer.
* Has read, understood, and signed the information consent letter.
* Has been diagnosed with dry eyes.
* Has reduced tear break up time (NITBUT) and/or reduced tear meniscus height (TMH), clinical sign of dry eye disease and contact lens discomfort or is symptomatic of dry eye.
* Is willing and able to follow instructions and maintain the appointment schedule.
* Has greater than 13 points on the OSDI.
* Has greater than 4 points on the Standardized Patient Evaluation of Eye Dryness (SPEED).

Exclusion Criteria:

A person will be excluded from the study if he/she:

* Is using any topical medications that will likely affect the study outcome.
* Has undergone any form of corneal surgery.
* Has any known allergies or sensitivity to the diagnostic pharmaceuticals or products, such as fluorescein, used in this study.
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye not related to the signs of dry eye.
* Has any clinically significant lid or conjunctival abnormalities and active neovascularization on the cornea.
* Anatomic variations of the conjunctiva that can impair proper scleral or soft contact lens wear/fitting
* Ocular pathology other than dry eye (e.g. glaucoma, macular degeneration) which may significantly impact visual function and assessment.
* Is participating in any other type of eye related clinical or research study.
* Has any active ocular infection and may require topical medications.
* Currently taking any systemic medication that may affect the study outcome.
* Is pregnant
* Has been diagnosed, recovered, or tested positive but asymptomatic with COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, FCOptom, Principal Investigator — University of Waterloo
Locations (1):
- School of Optometry & Vision Science, University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single site between April 2022 and October 2022. The first participant was enrolled on April 14, 2022 and the last participant was enrolled on October 25, 2022.
Pre-assignment Details: Of 30 enrolled participants, 28 met inclusion criteria and 25 were randomized to treatment.
Groups:
- Coated/Uncoated Scleral Lens: Participants wear first wear lenses coated with Hydra-PEG.
  Hydra-PEG: Zen™ RC scleral lenses (Hydra-PEG coated)
  Participants then wear uncoated (control) lenses.
  Uncoated: Zen™ RC scleral lenses (non-coated)
- Uncoated/Coated Scleral Lens: Participants wear first uncoated (control) lenses.
  Uncoated: Zen™ RC scleral lenses (non-coated
  Participants wear then wear lenses coated with Hydra-PEG.
  Hydra-PEG: Zen™ RC scleral lenses (Hydra-PEG coated)
Period: Overall Study
Arm/Group | Coated/Uncoated Scleral Lens | Uncoated/Coated Scleral Lens
Started | 12 | 13
Completed | 10 | 10
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: All suitable participants eligible to participate in the study.
Groups:
- Overall Group: All suitable participants eligible to take part in the study.
Arm/Group | Overall Group
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.79 (7.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 12
  Race: Caucasian | 8
  Race: African/Black | 2
  Race: Indian | 4
  Race: Arab | 2
Region of Enrollment [Number; unit: participants]
  Canada | 28

OUTCOME MEASURES:

1. Primary Outcome: Mean Corneal Thickness
Description: Mean corneal thickness as measured with Pentacam HR (µm)
Time Frame: At screening
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Coated/Uncoated Scleral Lens | Uncoated/Coated Scleral Lens
Number analyzed (Participants) | 12 | 13
microns | 570.54 (38.97) | 560.73 (31.48)
Statistical Analysis 1: Comparison: Coated/Uncoated Scleral Lens vs Uncoated/Coated Scleral Lens; Test type: Other; p = 0.25, t-test, 2 sided

2. Primary Outcome: Mean Corneal Thickness
Description: Mean corneal thickness as measured with Pentacam HR (µm)
Time Frame: After 4 weeks wear of coated lens
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Coated/Uncoated Scleral Lens | Uncoated/Coated Scleral Lens
Number analyzed (Participants) | 10 | 10
microns | 552.70 (26.96) | 559.85 (35.31)
Statistical Analysis 1: Comparison: Coated/Uncoated Scleral Lens vs Uncoated/Coated Scleral Lens; Test type: Other; p = 0.36, t-test, 2 sided

3. Primary Outcome: Mean Corneal Thickness
Description: Mean corneal thickness as measured with Pentacam HR (µm)
Time Frame: After 4 weeks wear of uncoated lens
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Coated Scleral Lens | Uncoated Scleral Lens
Number analyzed (Participants) | 10 | 10
microns | 556.91 (29.83) | 556.87 (29.92)
Statistical Analysis 1: Comparison: Coated Scleral Lens vs Uncoated Scleral Lens; Test type: Other; p = 1.0, t-test, 2 sided

4. Primary Outcome: Contact Lens Dry Eye Questionnaire (CLDEQ-8) Score
Description: The CLDEQ-8 is a validated questionnaire used to quantify symptoms experienced by the contact lenses (CLs) wearer. The participants were asked to respond to 8 questions about how their CLs performed over the preceding 2-week period. 4 questions (Eye discomfort, Eye dryness, Changeable blurry vision and Closing your eyes) answered on a scale of 0=Never to 4=Constantly; 3 questions about the end of wearing time (Discomfort, Dryness, Changeable blurry vision) answered on a scale of 0=Never have it to 5=Very Intense and 1 question (Removing your lenses) on a scale of 1=Never to 6=Several times a day for a total possible score of 1(best) to 37 (worst).
Time Frame: After 2 weeks of wear of coated lens
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coated/Uncoated Scleral Lens | Uncoated/Coated Scleral Lens
Number analyzed (Participants) | 10 | 10
score on a scale | 14.10 (7.92) | 20.30 (5.56)
Statistical Analysis 1: Comparison: Coated/Uncoated Scleral Lens vs Uncoated/Coated Scleral Lens; Test type: Other; p = 0.06, t-test, 2 sided

5. Primary Outcome: Contact Lens Dry Eye Questionnaire (CLDEQ-8) Score
Description: as for outcome 4
Time Frame: After 2 weeks of wear of uncoated lens
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coated/Uncoated Scleral Lens | Uncoated/Coated Scleral Lens
Number analyzed (Participants) | 10 | 10
score on a scale | 19.40 (7.34) | 17.20 (6.55)
Statistical Analysis 1: Comparison: Coated/Uncoated Scleral Lens vs Uncoated/Coated Scleral Lens; Test type: Other; p = 0.49, t-test, 2 sided

6. Primary Outcome: Contact Lens Dry Eye Questionnaire (CLDEQ-8) Score
Description: as for outcome 4
Time Frame: After 4 weeks of wear of coated lens
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coated/Uncoated Scleral Lens | Uncoated/Coated Scleral Lens
Number analyzed (Participants) | 10 | 10
score on a scale | 13.50 (7.07) | 19.50 (6.64)
Statistical Analysis 1: Comparison: Coated/Uncoated Scleral Lens vs Uncoated/Coated Scleral Lens; Test type: Other; p = 0.07, t-test, 2 sided

7. Primary Outcome: Contact Lens Dry Eye Questionnaire (CLDEQ-8) Score
Description: as for outcome 4
Time Frame: After 4 weeks of wear of uncoated lens
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coated/Uncoated Scleral Lens | Uncoated/Coated Scleral Lens
Number analyzed (Participants) | 10 | 10
score on a scale | 18.60 (7.99) | 15.10 (7.65)
Statistical Analysis 1: Comparison: Coated/Uncoated Scleral Lens vs Uncoated/Coated Scleral Lens; Test type: Other; p = 0.33, t-test, 2 sided

8. Primary Outcome: Tear Film Osmolarity
Description: Tear film osmolarity measures with a Tearlab Osmolarity System
Time Frame: At screening
Measure: Mean (Standard Deviation); unit: mOsm/l
Arm/Group | Coated/Uncoated Scleral Lens | Uncoated/Coated Scleral Lens
Number analyzed (Participants) | 12 | 13
mOsm/l | 313.29 (22.18) | 309.69 (16.32)
Statistical Analysis 1: Comparison: Coated/Uncoated Scleral Lens vs Uncoated/Coated Scleral Lens; Test type: Other; p = 0.65, t-test, 2 sided

9. Primary Outcome: Tear Film Osmolarity
Description: Tear film osmolarity measures with a Tearlab Osmolarity System
Time Frame: After 4 weeks of wear of uncoated lens
Measure: Mean (Standard Deviation); unit: mOsm/l
Arm/Group | Coated Scleral Lens | Uncoated Scleral Lens
Number analyzed (Participants) | 10 | 10
mOsm/l | 300.00 (12.87) | 306.05 (12.87)

10. Primary Outcome: Tear Film Osmolarity
Description: Tear film osmolarity measures with a Tearlab Osmolarity System
Time Frame: After 4 weeks of wear of coated lens
Measure: Mean (Standard Deviation); unit: mOsm/l
Arm/Group | Coated/Uncoated Scleral Lens | Uncoated/Coated Scleral Lens
Number analyzed (Participants) | 10 | 10
mOsm/l | 304.40 (8.48) | 303.90 (11.57)
Statistical Analysis 1: Comparison: Coated/Uncoated Scleral Lens vs Uncoated/Coated Scleral Lens; Test type: Other; p = 0.91, t-test, 2 sided

11. Primary Outcome: Contact Lens Impact on Quality of Life (CLIQ) Questionnaire Score
Description: This self-administered Contact Lens Impact on Quality of Life (CLIQ) questionnaire uses 28-item questions which are categorized into five main parameters: daily activities, eye symptoms, functional vision, psychometric properties, and refractive correction. Each question has a five-step response scale (none = 1; little = 2; moderate = 3; extreme = 4 and unable = 5). The responses are computed using the formula: CLIQperson measure = 34.41 × log (CLIQraw score/5 - CLIQraw score) + 26.69. This is then analyzed on a scale from 0 to 100, where higher scores indicate better QoL.
Time Frame: After 4 weeks of wear of uncoated lens
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coated/Uncoated Scleral Lens | Uncoated/Coated Scleral Lens
Number analyzed (Participants) | 10 | 10
score on a scale | 37.66 (13.37) | 39.67 (9.78)
Statistical Analysis 1: Comparison: Coated/Uncoated Scleral Lens vs Uncoated/Coated Scleral Lens; Test type: Other; p = 0.71, t-test, 2 sided

12. Primary Outcome: Contact Lens Impact on Quality of Life (CLIQ) Questionnaire Score
Description: as for outcome 11
Time Frame: After 4 weeks of wear of coated lens
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coated/Uncoated Scleral Lens | Uncoated/Coated Scleral Lens
Number analyzed (Participants) | 10 | 10
score on a scale | 40.70 (9.49) | 40.54 (11.31)
Statistical Analysis 1: Comparison: Coated/Uncoated Scleral Lens vs Uncoated/Coated Scleral Lens; Test type: Other; p = 0.97, t-test, 2 sided

13. Primary Outcome: Percentage of Participants With MMP-9 Inflammatory Marker in Tear Film
Description: Percentage of participants with a positive MMP-9 test, as measured by InflammaDry
Time Frame: At screening
Measure: Number; unit: percentage of participants
Arm/Group | Coated/Uncoated Scleral Lens | Uncoated/Coated Scleral Lens
Number analyzed (Participants) | 12 | 13
percentage of participants | 83.33 | 84.62
Statistical Analysis 1: Comparison: Coated/Uncoated Scleral Lens vs Uncoated/Coated Scleral Lens; Test type: Other; p = 0.75, Fisher Exact

14. Primary Outcome: Percentage of Participants With MMP-9 Inflammatory Marker in Tear Film
Description: Percentage of participants with a positive MMP-9 test, as measured by InflammaDry
Time Frame: After 4 weeks of wear of coated lens
Measure: Number; unit: percentage of participants
Arm/Group | Coated/Uncoated Scleral Lens | Uncoated/Coated Scleral Lens
Number analyzed (Participants) | 10 | 10
percentage of participants | 80 | 70
Statistical Analysis 1: Comparison: Coated/Uncoated Scleral Lens vs Uncoated/Coated Scleral Lens; Test type: Other; p = 0.59, Fisher Exact

15. Primary Outcome: Percentage of Participants With MMP-9 Inflammatory Marker in Tear Film
Description: Percentage of participants with a positive MMP-9 test, as measured by InflammaDry
Time Frame: After 4 weeks of wear of uncoated lens
Measure: Number; unit: percentage of participants
Arm/Group | Coated/Uncoated Scleral Lens | Uncoated/Coated Scleral Lens
Number analyzed (Participants) | 10 | 10
percentage of participants | 50 | 60
Statistical Analysis 1: Comparison: Coated/Uncoated Scleral Lens vs Uncoated/Coated Scleral Lens; Test type: Other; p = 0.69, Fisher Exact

ADVERSE EVENTS:
Time Frame: Maximum of three months
Description: Regular investigator assessment
Groups:
- Coated Scleral Lens: Participants wore lenses coated with Hydra-PEG.
  Hydra-PEG: Zen™ RC scleral lenses (Hydra-PEG coated)
- Uncoated Scleral Lens: Participants wore uncoated (control) lenses.
  Uncoated: Zen™ RC scleral lenses (non-coated)
Arm/Group | Coated Scleral Lens | Uncoated Scleral Lens
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT05079321/Prot_SAP_000.pdf